CLINICAL TRIAL: NCT05784675
Title: Impact of Serious Smartphone-based Game Use on Adult Performance of Basic Life Support Skills
Brief Title: Impact of Mobile Phone Application Use on Adult BLS
Acronym: MOBI-CPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nino Fijačko (Other)
Responsible Party: Sponsor-Investigator, Nino Fijačko, Principal Investigator, University Maribor
Organization: University Maribor (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MOBI-CPR game trial
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Mobile Phone Use; Stress; Knowledge, Attitudes, Practice
Keywords: basic life support; adult; mobile learning; stress; knowledge; skills; retention; home
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Cell Phone Use; Behavior

STUDY DESIGN:
Intervention Model Description: Balanced and randomized controlled cross-over within-subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOBI-CPR (Experimental): Participants use MOBI-CPR game at home environment.
  Interventions: Device: MOBI-CPR game
- No MOBI-CPR (No Intervention): Participants do not use MOBI-CPR game at home environment.

INTERVENTIONS:
Device: MOBI-CPR game — Participants use MOBI-CPR game at home environment.
  Arms: MOBI-CPR

SUMMARY:
The aim of the study is to investigate whether a serious smartphone game (called MOBI-CPR game) used in the home environment has an impact on the retention of adult basic life support knowledge and skills.

DETAILED DESCRIPTION:
The trial design will be randomized, controlled, cross-over study. Data will be collected between March and May 2023 at the Faculty of health science, University of Maribor. The consentience of nursing students will be collected. The Faculty of health science, University of Maribor already give permission for conducting this study. The goal will be to have around 100 nursing students in the study.

In the study a serious smartphone game called MOBI-CPR will be used. The MOBI-CPR game will be available at https://mobicpr.si/. The MOBI-CPR game will be install on the smartphone and will be used at home by nursing students with a goal to obtain adult basic life support knowledge and skills.

Before each nursing student will get MOBI-CPR game for home usage we will 1) measure acute stress, and 2) assess adult basic life support knowledge and skills.

For measuring acute stress the Empatica E4 watch will be used. Measuring will be perform in a quiet room without disruptions. When measuring acute stress each nursing student will be coloring the mandalas circles. Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).

For the knowledge part the online modified questionnaire (available in: https://www.1ka.si/d/en) the multiple choice questions will be used, and for the skills part the Resusci Anne QCPR QCPR manikin and Defibtech Trainer AED will be used. Each nursing student will be given the scenarios to read before the start of the assistance to the victim of a sudden cardiac arrest. The investigators will use a modified checklist to assess students' performance in adult basic life support.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students over eighteen years old
* Without training in adult basic life support or within the past six mounts
* Physically able to perform CPR
* Willingness to perform rescue breathing on a manikin
* A completed and signed consent form

Exclusion Criteria:

* Nursing student younger than 18 years old
* Undergone training on adult basic life support within the past six mounts
* Physically not able to perform CPR
* Do not want to perform rescue breathing on a manikin
* Do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Impact of the use of the MOBI-CPR game on the total score of theoretical adult basic life support knowledge | 2 weeks after baseline intervention
  Total score from the questionnaire (50 questions with multiple open answer, each right answer is 1 point) on the theoretical adult basic life support knowledge. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of theoretical adult basic life support knowledge | 4 weeks after baseline intervention
  Total score from the questionnaire (50 questions with multiple open answer, each right answer is 1 point) on the theoretical adult basic life support knowledge. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of theoretical adult basic life support knowledge | 6 mounts after baseline intervention
  Total score from the questionnaire (50 questions with multiple open answer, each right answer is 1 point) on the theoretical adult basic life support knowledge. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of theoretical adult basic life support knowledge | 1 year after baseline intervention
  Total score from the questionnaire (50 questions with multiple open answer, each right answer is 1 point) on the theoretical adult basic life support knowledge. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of theoretical adult basic life support knowledge | 3 years after baseline intervention
  Total score from the questionnaire (50 questions with multiple open answer, each right answer is 1 point) on the theoretical adult basic life support knowledge. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of practical adult basic life support skills | 2 weeks after baseline intervention
  Total score from the checklist (20 steps with correct or not correct assess of the adult basic life support, each right assess is 1 point) on the practical adult basic life support skills. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of practical adult basic life support skills | 4 weeks after baseline intervention
  Total score from the checklist (20 steps with correct or not correct assess of the adult basic life support, each right assess is 1 point) on the practical adult basic life support skills. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of practical adult basic life support skills | 6 mounts after baseline intervention
  Total score from the checklist (20 steps with correct or not correct assess of the adult basic life support, each right assess is 1 point) on the practical adult basic life support skills. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of practical adult basic life support skills | 1 year after baseline intervention
  Total score from the checklist (20 steps with correct or not correct assess of the adult basic life support, each right assess is 1 point) on the practical adult basic life support skills. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the total score of practical adult basic life support skills | 3 years after baseline intervention
  Total score from the checklist (20 steps with correct or not correct assess of the adult basic life support, each right assess is 1 point) on the practical adult basic life support skills. If the assessment score is over 70%, it indicates that the nursing student is successful.
Impact of the use of the MOBI-CPR game on the level of acute stress | 2 weeks after baseline intervention
  Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).
Impact of the use of the MOBI-CPR game on the level of acute stress | 4 weeks after baseline intervention
  Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).
Impact of the use of the MOBI-CPR game on the level of acute stress | 6 mounts after baseline intervention
  Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).
Impact of the use of the MOBI-CPR game on the level of acute stress | 1 year after baseline intervention
  Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).
Impact of the use of the MOBI-CPR game on the level of acute stress | 3 years after baseline intervention
  Level of acute stress measure by Empatica E4 watch (1-5 is non stress area, and 6-10 is stress area).

CONTACTS AND LOCATIONS:
Overall Officials: Nino Fijačko, Msc, Principal Investigator — University of Maribor, Faculty of Health Sciences
Locations (1):
- University of Maribor Faculty of health sciences, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez-Padilla J, Suthers F, Fernandez-Sola C, Granero-Molina J. Development and psychometric assessment of the Basic Resuscitation Skills Self-Efficacy Scale. Eur J Cardiovasc Nurs. 2016 Apr;15(3):e10-8. doi: 10.1177/1474515114562130. Epub 2014 Nov 24. PMID 25422522
- [Background] Papalexopoulou K, Chalkias A, Dontas I, Pliatsika P, Giannakakos C, Papapanagiotou P, Aggelina A, Moumouris T, Papadopoulos G, Xanthos T. Education and age affect skill acquisition and retention in lay rescuers after a European Resuscitation Council CPR/AED course. Heart Lung. 2014 Jan-Feb;43(1):66-71. doi: 10.1016/j.hrtlng.2013.09.008. Epub 2013 Oct 11. PMID 24246726
- [Derived] Fijacko N, Masterson Creber R, Metlicar S, Strnad M, Greif R, Stiglic G, Skok P. Effects of a Serious Smartphone Game on Nursing Students' Theoretical Knowledge and Practical Skills in Adult Basic Life Support: Randomized Wait List-Controlled Trial. JMIR Serious Games. 2024 Apr 5;12:e56037. doi: 10.2196/56037. PMID 38578690
- See also: Empatica E4 watch — https://www.empatica.com/
- See also: Software for questionnaire — https://www.1ka.si/d/en
- See also: Resusci Anne QCPR manikin — https://laerdal.com/distributors/products/simulation-training/resuscitation-training/resusci-anne-qcpr/
- See also: AED Defibtech Trainer AED — https://www.defibtech.com/products/aed-trainers/